CLINICAL TRIAL: NCT05835206
Title: A Randomized Controlled Trial to Further Microbiota Therapy for Antibiotic-Resistant Bacterial Colonization in Inpatients.
Brief Title: Further MT for Antibiotic-Resistant Bacterial Colonization in Inpatients
Acronym: FAIR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Woodworth, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00003613; 1U54CK000601-01 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Multi-drug Resistant Organism
Keywords: Carbapenem-resistant Enterobacteriaceae (CRE); Vancomycin-Resistant Enterococcus (VRE); Extended Spectrum Beta-Lactamase (ESBL); Multi-Drug Resistant (MDR) Acinetobacter; Multi-Drug Resistant (MDR) Pseudomonas
MeSH Terms: conditions — Pseudomonas Infections | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- microbiome therapeutic (Experimental): The study intervention is manufactured from a healthy screened donor as an investigational product (IP) and delivered via swallowed capsule after room reset of the patient's hospital room.
  Interventions: Drug: Microbiome Therapeutic
- Placebo (Placebo Comparator): The control arm will remain in routine contact precautions per standard of care, take placebo capsules, and have a room reset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Microbiome Therapeutic — Participants will receive a single course of study treatment (IP, Encapsulated Microbiota): Orally delivered, non-frozen, encapsulated investigational intestinal microbiota, consisting of 16 capsules. One dose (8 capsules) is administered daily (QD) for 2 days. The capsules are to be taken orally with water on an empty stomach. Each dose will be taken approximately every 24 hours, with a minimum of 12 hours from the previous dose to a maximum of 36 hours. Both doses must be completed within the stated 36 hours ±12 hours. Depending on the time of the first dose, dosing may occur over 3 calendar days.
  A second cycle will begin and a second treatment will be given if the participant is still MDRO positive on Day 14 of Cycle 1. If applicable, Cycle 2 will begin within 7 days of Day 14.
  Other Names: Intervention Group
  Arms: microbiome therapeutic
Drug: Placebo — Participants will receive a single course of study treatment (Color-matched placebo capsules containing microcrystalline cellulose (MCC) powder), consisting of 16 capsules. One dose (8 capsules) is administered daily (QD) for 2 days. The capsules are to be taken orally with water on an empty stomach. Each dose will be taken approximately every 24 hours, with a minimum of 12 hours from the previous dose to a maximum of 36 hours. Both doses must be completed within the stated 36 hours ±12 hours. Depending on the time of the first dose, dosing may occur over 3 calendar days.
  A second cycle will begin and a second treatment will be given if the participant is still MDRO positive on Day 14 of Cycle 1. If applicable, Cycle 2 will begin within 7 days of Day 14.
  Other Names: Control Group
  Arms: Placebo

SUMMARY:
The purpose of this study is to better understand the effectiveness and safety of microbiome therapies (MT) as a treatment for patients with Multidrug Resistant Organism (MDRO) colonization after an infection. Limited data from prior studies suggest that MT may be an effective treatment to reduce intestinal MDRO colonization Although shedding of MDROs from patients to their surrounding environment is a recognized pathway of transmission, the potential effect of MT on the transmission of MDRO to other patients in the hospital environment is unclear. This study will test the safety and efficacy of MT for this use in hospitalized patients. This study will also help design larger studies.

The MT may help reduce MDROs that colonize the gut. By reducing colonization before infections happen, this could help doctors avoid using "last resort" antibiotics that can have serious side effects like kidney damage. The reduction in MDROs after MT was originally identified in patients treated with MT for recurrent Clostridioides difficile (often called "C. diff") diarrhea. It has been shown that a type of MT called fecal microbiota transplant (FMT) can eliminate both C. difficile and other resistant bacteria.

DETAILED DESCRIPTION:
Antimicrobial resistance (AR) has been declared by the World Health Organization to be one of the greatest threats to global health. Every year, at least 2 million people are infected with antibiotic-resistant bacteria, and over 23,000 die from such infections.

This study aims to take initial steps to directly address these public health priorities and clinical threats of MDRO by estimating the safety of the IP in reducing patient-level intestinal MDRO colonization as well as the effect of the IP on environmental contamination. FAIR is a phase 2, randomized, placebo-controlled, double-blind, parallel, clinical trial of the IP for the treatment of MDRO colonization.

The hypothesis is that lyophilized human intestinal microbiota will safely and efficaciously reduce MDRO colonization. This is a randomized, controlled, clinical trial with two arms: a placebo arm and an intervention arm. The target population will include 40 adult inpatients with multi-drug resistant organisms (MDRO) colonization after infection. Target MDRO colonization is defined as a positive clinical microbiology bacterial culture and antibiotic susceptibility result that is consistent with one or more of the following: carbapenem-resistant Enterobacteriaceae (CRE), vancomycin-resistant Enterococcus spp (VRE), extended-spectrum β-lactamase (ESBL) producing Enterobacteriaceae, multidrug-resistant (MDR) Acinetobacter and/or MDR Pseudomonas

ELIGIBILITY:
Inclusion Criteria:

* Be able to (or have an available Legally Authorized Representative who is able to) understand and be willing to sign a written informed consent document.
* Be at least 18 years old at the time of consent.
* Be able and willing to comply with all study protocol requirements, including the ability to swallow capsules.
* Be colonized with a target MDRO (CRE, VRE, ESBL, MDR Acinetobacter, and/or MDR Pseudomonas) as detected by bacterial culture of stool or perianal/rectal swab.
* Be able and willing to discontinue systemic antibiotics at least one day prior to study Day 0 and for as long as medically able to do so throughout the study.
* Be willing to discontinue probiotics or other microbiota restoration therapies at least one day prior to study Day 0 and for the duration of study participation.
* The effects of the IP on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Be pregnant, breastfeeding, lactating, or planning a pregnancy during the study duration (through 4 weeks after the last dose of investigational product, or IP), if women of childbearing potential (WOCBP).
* Have known uncontrolled intercurrent illness(es) such as, but not limited to Symptomatic congestive heart failure, acute coronary syndrome, cardiac arrhythmia, untreated in situ colorectal cancer, toxic megacolon or ileus, use of medications that decrease GI motility and increase broncho-aspiration risk (e.g. loperamide, diphenoxylate/atropine, cholestyramine), or history of positive stool studies or cultures in the last 30 days for ova, parasites, Salmonella, Shigella, Campylobacter, or other enteropathogens other than those detected by screening MDRO stool cultures for inclusion.
* Have any other intercurrent acute illness that in the opinion of the investigator will preclude the subject from entering the study.
* Be on systemic antibiotics for any reason other than if the MDRO infection was recent or the potential participant is still taking antibiotics for target MDRO at the time of screening. If the latter, the participant must be able (in the opinion of their treating providers) to complete the planned antibiotic course by study Day -1.
* Have a compromised immune system, defined as AIDS with a cluster of differentiation 4 (CD4)+ T-cell count <200, history of documented absolute neutrophil count (ANC) <1,000 neutrophils/mL within 14 days of D0, active malignancy requiring intensive induction chemotherapy, radiotherapy, or biologic treatment within 2 months of enrollment or history of hematopoietic cell transplantation, either allogeneic or autologous in the last 1 year.
* Have a history of significant food allergy that led to anaphylaxis or hospitalization.
* Have a life expectancy of 24 weeks or less
* Have any condition that, in the opinion of the investigator, might interfere with study objectives or limit compliance with study requirements, including but not limited to known active intravenous drug or alcohol abuse, psychiatric illness, and/or social situation
* Participated in an investigational study that also meets one of the following criteria: Received an interventional agent (drug, device, or procedure) in the last 28 days or enrollment in any other interventional study for MDROs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in stool MDRO colony-forming unit (CFU) density | Day 0, day 14 of last cycle (each cycle is 14 days), and 28 weeks
  MDRO colony-forming unit (CFU) densities from quantitative stool cultures in placebo vs IP-treated participants.
Change in proportion of MDRO colonized participants after last treatment cycle with the investigational product (IP) | Day 0, day 14 of last cycle (each cycle is 14 days), and 28 weeks
  Proportion of stool cultures positive for any target MDRO will be compared in IP-treated vs placebo-treated participants.

SECONDARY OUTCOMES:
Estimate safety of the IP for MDRO colonization after infection | Day 0, day 7, day 14 of last cycle (each cycle is 14 days), and 28 weeks
  The frequency of adverse events from IP efficacy for reducing recurrent MDRO infection will be assessed by the frequency of MDRO infections at 24 weeks
Severity of adverse events caused by administration of the investigational product | Day 0, day 7, day 14 of last cycle (each cycle is 14 days), and 28 weeks
  Severity of adverse events after administration of MT will be graded as mild, moderate or severe, form the time of MT administration up to 24 weeks.
Estimate efficacy of the IP for reducing recurrent MDRO infection | Day 0, 24 weeks post Day 14 of last cycle (each cycle is 14 days)
  Efficacy will be measured by the frequency of MDRO infections from Day 0 of the first cycle until 24 weeks
Time to recurrent MDRO infection after IP administration | Day 0, 24 weeks post Day 14 of last cycle (each cycle is 14 days)
  Time to recurrent MDRO infection from Day 0 of first cycle censored at last final safety visit, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woodworth, MD, MSc, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Rehabilitation Hospital, Atlanta, Georgia
  - Emory University Clinical Research Network, Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Emory University at Wesley Woods Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The researchers will share all deidentified data included in the publication without restriction.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication
Access Criteria: Data will be uploaded to relevant repositories (e.g. National Center for Biotechnology Information (NCBI), Sequence Read Archive (SRA) for sequencing data and Dataverse or similar for clinical trial data)